CLINICAL TRIAL: NCT02149589
Title: Lung Imaging for Ventilatory Setting in ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: AZUREA group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHU-0192; 2013-A01756-39
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: ARDS
Keywords: ARDS; PEEP; Recruitment manoeuvres; Lung Morphology
MeSH Terms: interventions — Respiration, Artificial

ARMS (2):
- Focal ARDS (Experimental): In Focal ARDS prone position will be promote early, with low PEEP and moderate Vt.
  Interventions: Procedure: Mechanical ventilation
- non focal ARDS (Other): In non-Focal ARDS, Recruitment maneuvers, high PEEP and low V twill be used
  Interventions: Procedure: Mechanical ventilation

INTERVENTIONS:
Procedure: Mechanical ventilation

SUMMARY:
To compare in ARDS patients 2 ventilatory Strategies : One based on Lung Morphology (Focal versus non-Focal ARDS) versus ARDS networks Guidelines (PEEP based on FiO2). In Focal ARDS prone position will be promote early, with low PEEP and moderate Vt. In non-Focal ARDS, Recruitment maneuvers, high PEEP and low V twill be used.

The investigators made the hypothesis that ventilation according to Lung morphology my decrease mortality at D90.

DETAILED DESCRIPTION:
Early ARDS, less than 12 hours will be included. After Lung imaging, they will be randomized to a control group (PEEP/FiO2 according to ARDSnetwork tables) or an intervention arm. In this arm, mechanical ventilation will be set according to lung morphology. In patients with focal ARDS, prone position will be start quickly for at least 16 hours. After, A low PEEP and 8ml/kg of PBWwill be used. In non-focal ARDS, a recruitment maneuver followed by a high PEEP and a small tidal volume strategy will be used. In both arms, patients will be sedated and paralyzed during maximum 48 hours. As soon as PaO2/FiO2 > 200 mmHG, myorelaxant and sedation will be withdrawal. Pressure support ventilation will be used as soon as possible and weaning from ventilation will be checked everyday

ELIGIBILITY:
Inclusion Criteria:

* Man or female older than 18 years
* ARDS since less than 12 hours
* PaO2 / FiO2 < 200 avec une PEEP ≥ 5 (Berlin Moderate or severe)

Exclusion Criteria:

* brain injury with high ICP
* BMT Liver Cirrhosis Child C Pregnancy Burns Morbid obese patients (BMI > 40) Moribund

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Mortality rate | at day 90

SECONDARY OUTCOMES:
sRAGE & esRAGE plasmatic concentrations | at Day 0 Day 1 Day 2 Day 3 Day 4 Day 6 .
Quality of life | at Day 365

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CONSTANTIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Blanchard F, Godet T, Pons S, Kapandji N, Jabaudon M, Degos V, Borao L, Bougle A, Monsel A, Futier E, Constantin JM, James A. One-year patient outcomes based on lung morphology in acute respiratory distress syndrome: secondary analysis of LIVE trial. Crit Care. 2022 Jun 4;26(1):159. doi: 10.1186/s13054-022-04036-7. PMID 35659328
- [Derived] Constantin JM, Jabaudon M, Lefrant JY, Jaber S, Quenot JP, Langeron O, Ferrandiere M, Grelon F, Seguin P, Ichai C, Veber B, Souweine B, Uberti T, Lasocki S, Legay F, Leone M, Eisenmann N, Dahyot-Fizelier C, Dupont H, Asehnoune K, Sossou A, Chanques G, Muller L, Bazin JE, Monsel A, Borao L, Garcier JM, Rouby JJ, Pereira B, Futier E; AZUREA Network. Personalised mechanical ventilation tailored to lung morphology versus low positive end-expiratory pressure for patients with acute respiratory distress syndrome in France (the LIVE study): a multicentre, single-blind, randomised controlled trial. Lancet Respir Med. 2019 Oct;7(10):870-880. doi: 10.1016/S2213-2600(19)30138-9. Epub 2019 Aug 6. PMID 31399381
- [Derived] Jabaudon M, Godet T, Futier E, Bazin JE, Sapin V, Roszyk L, Pereira B, Constantin JM; AZUREA group. Rationale, study design and analysis plan of the lung imaging morphology for ventilator settings in acute respiratory distress syndrome study (LIVE study): Study protocol for a randomised controlled trial. Anaesth Crit Care Pain Med. 2017 Oct;36(5):301-306. doi: 10.1016/j.accpm.2017.02.006. Epub 2017 Mar 18. PMID 28323236